CLINICAL TRIAL: NCT02755688
Title: Catheter Ablation Versus Thoracoscopic Surgical Ablation in Long Standing Persistent Atrial Fibrillation (CASA-AF)
Acronym: CASA-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014CI005B
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Persistent Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; thoracoscopic surgical ablation; long standing persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracoscopic surgical ablation (Experimental): Pulmonary vein isolation, ganglionic plexi ablation, left atrial appendage exclusion
  Interventions: Procedure: Thoracoscopic Surgical ablation
- Catheter ablation (Active Comparator): Pulmonary vein isolation, linear lines
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Thoracoscopic Surgical ablation — Thoracoscopic approach to isolate pulmonary veins, ganglionic plexi ablation and left atrial appendage exclusion
  Arms: Thoracoscopic surgical ablation
Procedure: Catheter ablation — Ablation using contact force technology to isolate pulmonary veins and create linear lesions.
  Arms: Catheter ablation

SUMMARY:
Atrial fibrillation (AF) is the most common heart arrhythmia. Many people do not have symptoms and are not aware they have AF. Others may feel dizzy, short of breath, feel very tired and become aware of a fast and irregular heart beat (palpitations). The main complication of AF is an increased risk of stroke and incidence of heart failure. There are two key aspects of treatment for AF. The first is protection from stroke, treated with oral anticoagulants. Treatment of AF is either by controlling the rate (frequency of contraction) or controlling the rhythm (restoring regular contraction). Rate-control is generally employed first with an intent to reduce the rate at which the lower pumping chambers contract and improve their efficiency. Appropriate medication is used and with this treatment strategy it is accepted that AF will be present as the long term heart rhythm. If symptoms persist despite medication the preferred strategy is to restore sinus rhythm (SR) and regular contraction in all pumping chambers of the heart. This can be done with electric shock treatment (DC cardioversion) together with long-term tablet medication, or by a more definitive 'cauterisation' therapy (catheter or thoracoscopic surgical ablation). In this study the investigators will study patients with symptomatic long standing persistent AF (continuous AF for more than 1 year) who have tried and failed drug and/or electrical therapy. At present the investigators do not know what the best ablation technique is for treating symptomatic, long-standing persistent AF (LSPAF). Catheter ablation (CA) is the most widely available invasive treatment available for AF. Thoracoscopic surgical ablation (SA) is not widely available but our hospitals have the expertise to conduct this procedure. CA has been shown to achieve modest degrees of success in restoring normal SR with the caveat that most patients do require 'multiple' procedures (usually two or three). SA offers patients an alternative choice of therapy with a keyhole surgical thoracoscopic) approach. It may have a higher single procedure success rate although there is the potential for greater complication rates. The investigators aim to examine this in detail to help us understand which approach might be better for managing LSPAF.

DETAILED DESCRIPTION:
This is a multi-center randomised controlled study of catheter ablation compared with totally thoracoscopic surgical ablation.

The study population will be patients above the age of 18 with symptomatic long-standing persistent atrial fibrillation (≥1≤5 years) and good left ventricular function where at least one anti-arrhythmic drug (AAD) has failed, or where such drugs are contraindicated or not tolerated.

Subjects randomised to thoracoscopic Surgical Ablation will undergo minimally invasive, thoracoscopically assisted, surgical ablation to isolate the pulmonary veins (PVI) using a radiofrequency (RF) clamp device. Posterior wall will be isolated in a box fashion with cool rail bipolar RF device. This will include ganglionated plexi ablation +/- LAA excision/exclusion.

Catheter Ablation Group Patients will undergo pulmonary vein isolation and linear ablations in the left and right atrium.

There will be a 3 month blanking period and symptomatic atrial arrhythmia may have catheter ablation during the period of 12 month follow up. The primary end point of the study will be assessed by continuous cardiac recording through an internal loop recorder that will be inserted at the end of the index procedure. The analysis and reporting of the recordings will be performed by a blinded core lab.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 yrs.
2. LSPAF (> 12 months' duration)
3. EHRA>2
4. Left ventricular ejection fraction ≥ 40%
5. Suitable for either ablation procedure

Exclusion Criteria:

1. Left sided valvular heart disease with severity greater than mild
2. Contraindication to anticoagulation
3. Thrombus in the left atrium despite anticoagulation in therapeutic range
4. Cerebrovascular accident within the previous 6 months
5. Previous thoracic or cardiac surgery (including surgical interventions for AF)
6. Prior left atrial catheter ablation for AF
7. Unable to provide informed written consent
8. Active malignancy, another severe concomitant condition or presence of implanted intracardiac devices that would preclude patient undergoing study specific procedures
9. Pregnant or breast-feeding, or women of childbearing age not using a reliable contraceptive method.
10. Implanted non MRI compatible cardiac devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06; Primary Completion 2019-10-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias (>30 seconds) after a single procedure without anti-arrhythmic drugs (AADs) within 12 months measured by internal loop recorder | 12 months
  All patients will have internal loop recorder inserted after the completion of the procedure and the data will be analysed by a blinded core lab. 3 months of the blanking period will not be counted as accepted by EHRA / HRS committee. The definition of atrial arrhythmias is equal to or greater than 30 seconds of atrial tachycardia or atrial fibrillation as mentioned in EHRA / HRS consensus statement 2012.

SECONDARY OUTCOMES:
Intervention-related major complication rate defined as permanent injury or death, requires unplanned intervention for treatment, or prolongs or requires unplanned hospitalization for more than 48 hours | 12 months
Clinical success from the arrhythmia interventions - defined as a 75% or greater reduction of AF burden with or without AADs. | 12 months
Freedom from atrial arrhythmia, after multiple procedures without AADs | 12 months
  Measured by internal loop recorder and analysed by blinded core lab.
Changes in atrial anatomy and function following ablation as assessed by echocardiography using tissue Doppler and strain | 12 months
Changes in atrial anatomy and atrial fibrosis following ablation as assessed by cardiac MRI | 12 months
Effects of the arrhythmia interventions on the patients' symptoms by Change in AF symptom score (EHRA score) | 12 months
Effects of the arrhythmia interventions on the quality of life as assessed by change in quality of life assessments (EQ5D) | 12 months
Effects of the arrhythmia interventions on the quality of life as assessed by change in quality of life assessments (AFEQT) | 12 months
Quality Adjusted Life Years (QALYs) accrued during follow up | 12 months
Cost-effectiveness (Incremental Cost per QALY gained) for surgical ablation compared with CA estimated | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wong, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton and Harefield Hospital NHS Trusts, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan HR, Yakupoglu HY, Kralj-Hans I, Haldar S, Bahrami T, Clague J, De Souza A, Hussain W, Jarman J, Jones DG, Salukhe T, Markides V, Gupta D, Khattar R, Wong T; CASA AF Investigators. Left Atrial Function Predicts Atrial Arrhythmia Recurrence Following Ablation of Long-Standing Persistent Atrial Fibrillation. Circ Cardiovasc Imaging. 2023 Jun;16(6):e015352. doi: 10.1161/CIRCIMAGING.123.015352. Epub 2023 Jun 8. PMID 37288553
- [Derived] Haldar S, Khan HR, Boyalla V, Kralj-Hans I, Jones S, Lord J, Onyimadu O, Satishkumar A, Bahrami T, De Souza A, Clague JR, Francis DP, Hussain W, Jarman JW, Jones DG, Chen Z, Mediratta N, Hyde J, Lewis M, Mohiaddin R, Salukhe TV, Murphy C, Kelly J, Khattar RS, Toff WD, Markides V, McCready J, Gupta D, Wong T. Catheter ablation vs. thoracoscopic surgical ablation in long-standing persistent atrial fibrillation: CASA-AF randomized controlled trial. Eur Heart J. 2020 Dec 14;41(47):4471-4480. doi: 10.1093/eurheartj/ehaa658. PMID 32860414